CLINICAL TRIAL: NCT00964158
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (GSK2340272A) in Children Aged 3 to 17 Years
Brief Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (H1N1) (GSK2340272A)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 113528
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: Pandemic influenza vaccine GSK2340272A

INTERVENTIONS:
Biological: Pandemic influenza vaccine GSK2340272A — Two primary intramuscular (IM) injections and a booster IM injection

SUMMARY:
This trial is designed to assess the safety and immunogenicity of a prime-boost schedule of GSK Biologicals' investigational vaccine GSK2340272A in children aged between 3 and 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Children, male or female, aged between 3 and 17 years at the time of the first study vaccination.
* Written informed consent obtained from the subject parent(s) or LAR(s) of the subject. Assent obtained from the subject when applicable.
* Healthy children as established by medical history and clinical examination when entering into the study.
* Parent/LAR with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Clinically or virologically confirmed influenza infection within six months preceding the study start.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Previous administration of any H1N1 A/California-like vaccine.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* If the subject is female and if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.
* Any known or suspected allergy to any constituent of influenza vaccines;a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* Known use of an analgesic or antipyretic medication within 12 hours prior to first vaccination.
* Child in Care.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2009-09-10; Primary Completion 2010-11-27 (Actual); Study Completion 2010-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Spain (5):
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Garcia-Sicilia J, Aristegui J, Omenaca F, Carmona A, Tejedor JC, Merino JM, Garcia-Corbeira P, Walravens K, Bambure V, Moris P, Caplanusi A, Gillard P, Dieussaert I. Safety and persistence of the humoral and cellular immune responses induced by 2 doses of an AS03-adjuvanted A(H1N1)pdm09 pandemic influenza vaccine administered to infants, children and adolescents: Two open, uncontrolled studies. Hum Vaccin Immunother. 2015;11(10):2359-69. doi: 10.1080/21645515.2015.1063754. PMID 26176592
- [Derived] Garcia-Sicilia J, Gillard P, Carmona A, Tejedor JC, Aristegui J, Merino JM, Behre U, Caplanusi A, Vaman T, Dieussaert I. Immunogenicity and safety of AS03-adjuvanted H1N1 pandemic vaccines in children and adolescents. Vaccine. 2011 Jun 10;29(26):4353-61. doi: 10.1016/j.vaccine.2011.04.011. Epub 2011 Apr 17. PMID 21504774
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113528 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- GSK2340272A (3-5Y) Group: Healthy male or female children between 3 to 5 years of age (3-5Y), who received 2 primary doses of GSK2340272A vaccine according to a 0, 21-day schedule, administered intramuscularly in the deltoid region of the arm.
- GSK2340272A (6-9Y) Group: Healthy male or female children between 6 to 9 years of age (6-9Y), who received 2 primary doses of GSK2340272A vaccine according to a 0, 21-day schedule, administered intramuscularly in the deltoid region of the arm.
- GSK2340272A (10-17Y) Group: Healthy male or female children between 10 to 17 years of age (10-17Y), who received 2 primary doses of GSK2340272A vaccine according to a 0, 21-day schedule, administered intramuscularly in the deltoid region of the arm.
Period: Overall Study
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Started | 53 | 57 | 100
Completed | 53 | 56 | 92
Not Completed | 0 | 1 | 8
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group | Total
Number analyzed (Participants) | 53 | 57 | 100 | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.5 (0.7) | 7.5 (1.18) | 13.3 (2.23) | 9.25 (4.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 61 | 117
  Male | 22 | 32 | 39 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian - East Asian heritage | 0 | 1 | 0 | 1
  Geographic ancestry: White - Caucasian/European heritage | 53 | 56 | 99 | 208
  Geographic ancestry: Unspecified | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Haemagglutination-inhibition (HI) Antibody Concentrations Above the Cut-off Value
Description: The seropositivity cut-off value of the assay was equal to or above (≥) 1:10 in the sera of subjects seronegative before vaccination. The flu strain assessed was A/California/7/2009 (H1N1)v-like (Flu A/CAL/7/09).
Time Frame: At Day 0
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 2 doses were taken and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the second vaccine dose given at Day 21.
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A Group: Healthy male or female children between 3 to 17 years of age, who received 2 primary doses of GSK2340272A vaccine according to a 0, 21-day schedule, administered intramuscularly in the deltoid region of the arm.
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 198
Participants | 40

2. Primary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: The seropositivity cut-off value of the assay was ≥ 1:10 in the sera of subjects seronegative before vaccination. The flu strain assesssed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 194
Participants | 194

3. Primary Outcome: Titers for Serum HI Antibodies
Description: Antibody titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:10. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects for whom 2 doses were taken and assay results were available for antibodies against H1N1 antigen for the blood sample taken 21 days after the second vaccine dose given at Day 21.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 198
Titers | 7.4 [6.4 to 8.5]

4. Primary Outcome: Titers for Serum HI Antibodies
Description: as for outcome 3
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 194
Titers | 1538.5 [1419.0 to 1668.2]

5. Primary Outcome: Number of Seroconverted (SCR) Subjects in Terms of HI Antibodies
Description: A seroconverted subject was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 prior to vaccination], antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), at least a 4-fold increase in post-vaccination titer. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 194
Participants | 191

6. Primary Outcome: Number of Seroprotected (SPR) Subjects in Terms of HI Antibodies
Description: Seroprotection was defined as the percentage of subjects with a serum HI titer ≥ 1:40, that usually is accepted as indicating protection. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 194
Participants | 194

7. Primary Outcome: Seroconversion Factor (SCF) for HI Antibody Titers
Description: Seroconversion factor was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A Group
Number analyzed (Participants) | 194
Fold increase | 208.5 [179.0 to 242.9]

8. Secondary Outcome: Number of Subjects With HI Antibody Concentrations Above the Cut-off Value
Description: as for outcome 2
Time Frame: At Days 0, 21, 42 and at Month 12
Population: The analysis was performed on the ATP cohort for persistence at Month 12, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against the study vaccine antigen component at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 42 | 50 | 87
Participants
  Flu A/CAL/7/09, Day 0 | 0 | 6 | 22
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 41 | 50 | 87
  Flu A/CAL/7/09, Day 21 | 41 | 50 | 87
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 41 | 49 | 83
  Flu A/CAL/7/09, Day 42 | 41 | 49 | 83
  Flu A/CAL/7/09, Month 12 | 42 | 50 | 87

9. Secondary Outcome: Titers for Serum HI Antibodies
Description: as for outcome 3
Time Frame: At Days 0, 21, 42 and at Month 12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 42 | 50 | 87
Titers
  Flu A/CAL/7/09, Day 0 | 5.0 [5.0 to 5.0] | 6.3 [5.2 to 7.7] | 8.9 [6.9 to 11.3]
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 41 | 50 | 87
  Flu A/CAL/7/09, Day 21 | 168.3 [140.5 to 201.6] | 284.4 [218.3 to 370.5] | 547.9 [457.1 to 656.8]
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 41 | 49 | 83
  Flu A/CAL/7/09, Day 42 | 1581.1 [1365.7 to 1830.6] | 964.6 [847.4 to 1098.0] | 1008.9 [881.3 to 1155.0]
  Flu A/CAL/7/09, Month 12 | 123.9 [102.8 to 149.3] | 106.3 [88.6 to 127.5] | 251.0 [206.6 to 304.9]

10. Secondary Outcome: Number of Seroconverted (SCR) Subjects in Terms of HI Antibodies
Description: A seroconverted subject was defined as: For initially seronegative subjects [antibody titer below (<) 1:10 prior to vaccination], antibody titer ≥ 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:10 prior to vaccination), at least a 4-fold increase in post-vaccination antibody titer. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Days 21, 42 and at Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 42 | 50 | 87
Participants
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 41 | 50 | 87
  Flu A/CAL/7/09, Day 21 | 41 | 50 | 85
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 41 | 49 | 83
  Flu A/CAL/7/09, Day 42 | 41 | 49 | 80
  Flu A/CAL/7/09, Month 12 | 42 | 48 | 82

11. Secondary Outcome: Number of Seroprotected Subjects in Terms of HI Antibodies
Description: as for outcome 6
Time Frame: At Days 0, 21, 42 and at Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 42 | 50 | 87
Participants
  Flu A/CAL/7/09, Day 0 | 0 | 3 | 12
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 41 | 50 | 87
  Flu A/CAL/7/09, Day 21 | 41 | 50 | 87
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 41 | 49 | 83
  Flu A/CAL/7/09, Day 42 | 41 | 49 | 83
  Flu A/CAL/7/09, Month 12 | 42 | 49 | 87

12. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibody Titers
Description: as for outcome 7
Time Frame: At Days 21, 42 and at Month 12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 42 | 50 | 87
Fold increase
  Flu A/CAL/7/09, Day 21: number analyzed (Participants) | 41 | 50 | 87
  Flu A/CAL/7/09, Day 21 | 33.7 [28.1 to 40.3] | 44.9 [36.0 to 56.1] | 61.8 [48.4 to 78.8]
  Flu A/CAL/7/09, Day 42: number analyzed (Participants) | 41 | 49 | 83
  Flu A/CAL/7/09, Day 42 | 316.2 [273.1 to 366.1] | 151.7 [123.4 to 186.5] | 119.8 [92.3 to 155.4]
  Flu A/CAL/7/09, Month 12 | 24.8 [20.6 to 29.9] | 16.8 [13.8 to 20.5] | 28.3 [22.2 to 36.1]

13. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: The seropositivity cut-off value of the assay was ≥ 1:8 in the sera of subjects seronegative before vaccination. The flu strain assesssed was Flu A/Neth/602/09.
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 32 | 37 | 30
Participants
  Flu A/Neth/602/09, Day 0 | 1 | 6 | 3
  Flu A/Neth/602/09, Day 21 | 31 | 37 | 30
  Flu A/Neth/602/09, Day 42: number analyzed (Participants) | 29 | 37 | 29
  Flu A/Neth/602/09, Day 42 | 29 | 37 | 29

14. Secondary Outcome: Titers for Serum Neutralizing Antibodies
Description: Antibody titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:8. The flu strain assessed was A/Netherlands/602/2009 (H1N1)v-like (Flu A/Neth/602/09).
Time Frame: At Days 0, 21 and 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 32 | 37 | 30
Titers
  Flu A/Neth/602/09, Day 0 | 4.1 [3.9 to 4.4] | 6.1 [4.2 to 8.8] | 5.3 [3.6 to 7.9]
  Flu A/Neth/602/09, Day 21 | 60.2 [42.4 to 85.5] | 149.0 [80.7 to 275.0] | 113.0 [71.5 to 178.8]
  Flu A/Neth/602/09, Day 42: number analyzed (Participants) | 29 | 37 | 29
  Flu A/Neth/602/09, Day 42 | 1277.4 [895.1 to 1822.9] | 751.0 [491.0 to 1148.6] | 553.4 [388.4 to 788.4]

15. Secondary Outcome: Number of Subjects With Neutralizing Antibody Concentrations Above the Cut-off Value
Description: as for outcome 13
Time Frame: At Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 25 | 32 | 28
Participants | 25 | 32 | 28

16. Secondary Outcome: Titers for Serum Neutralizing Antibodies
Description: Antibody titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was ≥ 1:8. The flu strain assessed was Flu A/Neth/602/09.
Time Frame: At Month 12
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 25 | 32 | 28
Titers | 269.1 [198.9 to 363.9] | 168.4 [121.0 to 234.4] | 118.1 [85.6 to 163.0]

17. Secondary Outcome: Number of Seroconverted (SCR) Subjects in Terms of H1N1 Neutralizing Antibodies
Description: A seroconverted subject was defined as: For initially seronegative subjects, antibody titer ≥ 1:32 after vaccination; For initially seropositive subjects, at least a 4-fold increase in post-vaccination titer. The flu strain assessed was Flu A/Neth/602/09.
Time Frame: At Days 21 and 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 32 | 37 | 30
Participants
  Flu A/Neth/602/09, Day 21 | 26 | 32 | 26
  Flu A/Neth/602/09, Day 42: number analyzed (Participants) | 29 | 37 | 29
  Flu A/Neth/602/09, Day 42 | 29 | 37 | 29

18. Secondary Outcome: Number of Seroconverted (SCR) Subjects in Terms of H1N1 Neutralizing Antibodies
Description: as for outcome 17
Time Frame: At Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 24 | 31 | 28
Participants | 24 | 30 | 25

19. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 98
Participants
  Any Pain, Dose 1 | 40 | 54 | 91
  Grade 3 Pain, Dose 1 | 2 | 3 | 8
  Any Redness, Dose 1 | 15 | 14 | 21
  Grade 3 Redness, Dose 1 | 0 | 2 | 6
  Any Swelling, Dose 1 | 18 | 16 | 41
  Grade 3 Swelling, Dose 1 | 1 | 3 | 6
  Any Pain, Dose 2: number analyzed (Participants) | 52 | 57 | 93
  Any Pain, Dose 2 | 44 | 55 | 90
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 52 | 57 | 93
  Grade 3 Pain, Dose 2 | 5 | 8 | 12
  Any Redness, Dose 2: number analyzed (Participants) | 52 | 57 | 93
  Any Redness, Dose 2 | 18 | 19 | 26
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 52 | 57 | 93
  Grade 3 Redness, Dose 2 | 4 | 2 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 52 | 57 | 93
  Any Swelling, Dose 2 | 16 | 26 | 50
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 52 | 57 | 93
  Grade 3 Swelling, Dose 2 | 2 | 1 | 2
  Any Pain, Across doses | 47 | 56 | 95
  Grade 3 Pain, Across doses | 7 | 8 | 16
  Any Redness, Across doses | 22 | 22 | 33
  Grade 3 Redness, Across doses | 4 | 4 | 6
  Any Swelling, Across doses | 25 | 30 | 60
  Grade 3 Swelling, Across doses | 3 | 4 | 6

20. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were diarrhea, drowsiness, irritability, loss of appetite, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group
Number analyzed (Participants) | 53
Participants
  Any Diarrhea, Dose 1 | 2
  Grade 3 Diarrhea, Dose 1 | 0
  Related Diarrhea, Dose 1 | 1
  Any Drowsiness, Dose 1 | 11
  Grade 3 Drowsiness, Dose 1 | 0
  Related Drowsiness, Dose 1 | 8
  Any Irritability, Dose 1 | 14
  Grade 3 Irritability, Dose 1 | 0
  Related Irritability, Dose 1 | 10
  Any Loss of appetite, Dose 1 | 14
  Grade 3 Loss of appetite, Dose 1 | 0
  Related Loss of appetite, Dose 1 | 8
  Any Shivering, Dose 1 | 5
  Grade 3 Shivering, Dose 1 | 0
  Related Shivering, Dose 1 | 2
  Any Sweating, Dose 1 | 4
  Grade 3 Sweating, Dose 1 | 0
  Related Sweating, Dose 1 | 1
  Any Temperature, Dose 1 | 14
  Grade 3 Temperature, Dose 1 | 1
  Related Temperature, Dose 1 | 8
  Any Diarrhea, Dose 2: number analyzed (Participants) | 52
  Any Diarrhea, Dose 2 | 6
  Grade 3 Diarrhea, Dose 2: number analyzed (Participants) | 52
  Grade 3 Diarrhea, Dose 2 | 0
  Related Diarrhea, Dose 2: number analyzed (Participants) | 52
  Related Diarrhea, Dose 2 | 3
  Any Drowsiness, Dose 2: number analyzed (Participants) | 52
  Any Drowsiness, Dose 2 | 17
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 52
  Grade 3 Drowsiness, Dose 2 | 2
  Related Drowsiness, Dose 2: number analyzed (Participants) | 52
  Related Drowsiness, Dose 2 | 15
  Any Irritability, Dose 2: number analyzed (Participants) | 52
  Any Irritability, Dose 2 | 15
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 52
  Grade 3 Irritability, Dose 2 | 3
  Related Irritability, Dose 2: number analyzed (Participants) | 52
  Related Irritability, Dose 2 | 14
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 52
  Any Loss of appetite, Dose 2 | 21
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 52
  Grade 3 Loss of appetite, Dose 2 | 3
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 52
  Related Loss of appetite, Dose 2 | 17
  Any Shivering, Dose 2: number analyzed (Participants) | 52
  Any Shivering, Dose 2 | 6
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 52
  Grade 3 Shivering, Dose 2 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 52
  Related Shivering, Dose 2 | 5
  Any Sweating, Dose 2: number analyzed (Participants) | 52
  Any Sweating, Dose 2 | 6
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 52
  Grade 3 Sweating, Dose 2 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 52
  Related Sweating, Dose 2 | 4
  Any Temperature, Dose 2: number analyzed (Participants) | 52
  Any Temperature, Dose 2 | 26
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 52
  Grade 3 Temperature, Dose 2 | 2
  Related Temperature, Dose 2: number analyzed (Participants) | 52
  Related Temperature, Dose 2 | 23
  Any Diarrhea, Across doses | 8
  Grade 3 Diarrhea, Across doses | 0
  Related Diarrhea, Across doses | 4
  Any Drowsiness, Across doses | 22
  Grade 3 Drowsiness, Across doses | 2
  Related Drowsiness, Across doses | 19
  Any Irritability, Across doses | 21
  Grade 3 Irritability, Across doses | 3
  Related Irritability, Across doses | 19
  Any Loss of appetite, Across doses | 28
  Grade 3 Loss of appetite, Across doses | 3
  Related Loss of appetite, Across doses | 21
  Any Shivering, Across doses | 11
  Grade 3 Shivering, Across doses | 1
  Related Shivering, Across doses | 7
  Any Sweating, Across doses | 10
  Grade 3 Sweating, Across doses | 0
  Related Sweating, Across doses | 5
  Any Temperature, Across doses | 33
  Grade 3 Temperature, Across doses | 3
  Related Temperature, Across doses | 26

21. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal, headache, myalgia, shivering and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 57 | 98
Participants
  Any Arthralgia, Dose 1 | 9 | 26
  Grade 3 Arthralgia, Dose 1 | 0 | 1
  Related Arthralgia, Dose 1 | 8 | 26
  Any Fatigue, Dose 1 | 21 | 44
  Grade 3 Fatigue, Dose 1 | 1 | 4
  Related Fatigue, Dose 1 | 20 | 40
  Any Gastrointestinal, Dose 1 | 13 | 12
  Grade 3 Gastrointestinal, Dose 1 | 2 | 1
  Related Gastrointestinal, Dose 1 | 9 | 6
  Any Headache, Dose 1 | 25 | 48
  Grade 3 Headache, Dose 1 | 2 | 3
  Related Headache, Dose 1 | 24 | 41
  Any Myalgia, Dose 1 | 15 | 35
  Grade 3 Myalgia, Dose 1 | 2 | 2
  Related Myalgia, Dose 1 | 13 | 34
  Any Shivering, Dose 1 | 7 | 19
  Grade 3 Shivering, Dose 1 | 0 | 0
  Related Shivering, Dose 1 | 4 | 14
  Any Sweating, Dose 1 | 2 | 8
  Grade 3 Sweating, Dose 1 | 0 | 0
  Related Sweating, Dose 1 | 1 | 5
  Any Temperature, Dose 1 | 13 | 17
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 10 | 15
  Any Arthralgia, Dose 2: number analyzed (Participants) | 57 | 93
  Any Arthralgia, Dose 2 | 13 | 34
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Arthralgia, Dose 2 | 1 | 1
  Related Arthralgia, Dose 2: number analyzed (Participants) | 57 | 93
  Related Arthralgia, Dose 2 | 13 | 32
  Any Fatigue, Dose 2: number analyzed (Participants) | 57 | 93
  Any Fatigue, Dose 2 | 29 | 50
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Fatigue, Dose 2 | 3 | 5
  Related Fatigue, Dose 2: number analyzed (Participants) | 57 | 93
  Related Fatigue, Dose 2 | 28 | 48
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 57 | 93
  Any Gastrointestinal, Dose 2 | 9 | 10
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 57 | 93
  Related Gastrointestinal, Dose 2 | 8 | 6
  Any Headache, Dose 2: number analyzed (Participants) | 57 | 93
  Any Headache, Dose 2 | 26 | 51
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Headache, Dose 2 | 4 | 5
  Related Headache, Dose 2: number analyzed (Participants) | 57 | 93
  Related Headache, Dose 2 | 26 | 50
  Any Myalgia, Dose 2: number analyzed (Participants) | 57 | 93
  Any Myalgia, Dose 2 | 16 | 47
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Myalgia, Dose 2 | 1 | 2
  Related Myalgia, Dose 2: number analyzed (Participants) | 57 | 93
  Related Myalgia, Dose 2 | 16 | 44
  Any Shivering, Dose 2: number analyzed (Participants) | 57 | 93
  Any Shivering, Dose 2 | 14 | 27
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Shivering, Dose 2 | 0 | 1
  Related Shivering, Dose 2: number analyzed (Participants) | 57 | 93
  Related Shivering, Dose 2 | 13 | 25
  Any Sweating, Dose 2: number analyzed (Participants) | 57 | 93
  Any Sweating, Dose 2 | 7 | 8
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Sweating, Dose 2 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 57 | 93
  Related Sweating, Dose 2 | 4 | 7
  Any Temperature, Dose 2: number analyzed (Participants) | 57 | 93
  Any Temperature, Dose 2 | 20 | 23
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 57 | 93
  Grade 3 Temperature, Dose 2 | 1 | 1
  Related Temperature, Dose 2: number analyzed (Participants) | 57 | 93
  Related Temperature, Dose 2 | 19 | 16
  Any Arthralgia, Across doses | 20 | 44
  Grade 3 Arthralgia, Across doses | 1 | 2
  Related Arthralgia, Across doses | 19 | 43
  Any Fatigue, Across doses | 35 | 63
  Grade 3 Fatigue, Across doses | 4 | 9
  Related Fatigue, Across doses | 34 | 59
  Any Gastrointestinal, Across doses | 17 | 16
  Grade 3 Gastrointestinal, Across doses | 2 | 1
  Related Gastrointestinal, Across doses | 14 | 10
  Any Headache, Across doses | 34 | 70
  Grade 3 Headache, Across doses | 5 | 6
  Related Headache, Across doses | 34 | 64
  Any Myalgia, Across doses | 23 | 56
  Grade 3 Myalgia, Across doses | 2 | 4
  Related Myalgia, Across doses | 21 | 53
  Any Shivering, Across doses | 19 | 38
  Grade 3 Shivering, Across doses | 0 | 1
  Related Shivering, Across doses | 15 | 33
  Any Sweating, Across doses | 9 | 14
  Grade 3 Sweating, Across doses | 0 | 0
  Related Sweating, Across doses | 5 | 11
  Any Temperature, Across doses | 27 | 33
  Grade 3 Temperature, Across doses | 1 | 1
  Related Temperature, Across doses | 23 | 25

22. Secondary Outcome: Number of Subjects With Any Medically-attended Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 100
Participants | 36 | 21 | 33

23. Secondary Outcome: Number of Subjects With Any Adverse Events of Specific Interest (AESIs), Including Potential Immune-mediated Disease (pIMDs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 100
Participants | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects With Normal or Abnormal Biochemical Levels
Description: Among biochemical parameters assessed were alanine aminotransferase [ALAT], aspartate aminotransferase [ASAT], bilirubin [BILI], creatinine [CREA] and blood urea nitrogen [BUN]. Levels of biochemical parameters assessed in terms of normal laboratory values were - unknown, below, within and above.
Time Frame: At Days 0, 21 and 42
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 97
Participants
  ALAT, Day 0: number analyzed (Participants) | 30 | 38 | 59
  ALAT, Day 0: Unknown | 0 | 0 | 0
  ALAT, Day 0: Below | 0 | 0 | 0
  ALAT, Day 0: Within | 30 | 38 | 59
  ALAT, Day 0: Above | 0 | 0 | 0
  ALAT, Day 21: Unknown | 1 | 0 | 2
  ALAT, Day 21: Below | 0 | 0 | 0
  ALAT, Day 21: Within | 52 | 57 | 94
  ALAT, Day 21: Above | 0 | 0 | 1
  ALAT, Day 42: number analyzed (Participants) | 52 | 56 | 93
  ALAT, Day 42: Unknown | 2 | 1 | 0
  ALAT, Day 42: Below | 0 | 0 | 0
  ALAT, Day 42: Within | 50 | 55 | 91
  ALAT, Day 42: Above | 0 | 0 | 2
  ASAT, Day 0: number analyzed (Participants) | 30 | 38 | 59
  ASAT, Day 0: Unknown | 0 | 0 | 0
  ASAT, Day 0: Below | 0 | 0 | 0
  ASAT, Day 0: Within | 28 | 38 | 58
  ASAT, Day 0: Above | 2 | 0 | 1
  ASAT, Day 21: Unknown | 2 | 1 | 2
  ASAT, Day 21: Below | 0 | 0 | 0
  ASAT, Day 21: Within | 50 | 56 | 94
  ASAT, Day 21: Above | 1 | 0 | 1
  ASAT, Day 42: number analyzed (Participants) | 52 | 56 | 93
  ASAT, Day 42: Unknown | 2 | 1 | 0
  ASAT, Day 42: Below | 0 | 0 | 0
  ASAT, Day 42: Within | 50 | 55 | 91
  ASAT, Day 42: Above | 0 | 0 | 2
  BILI, Day 0: number analyzed (Participants) | 30 | 38 | 59
  BILI, Day 0: Unknown | 0 | 0 | 0
  BILI, Day 0: Below | 0 | 0 | 0
  BILI, Day 0: Within | 30 | 38 | 57
  BILI, Day 0: Above | 0 | 0 | 2
  BILI, Day 21: Unknown | 1 | 0 | 2
  BILI, Day 21: Below | 0 | 0 | 0
  BILI, Day 21: Within | 52 | 57 | 90
  BILI, Day 21: Above | 0 | 0 | 5
  BILI, Day 42: number analyzed (Participants) | 52 | 56 | 93
  BILI, Day 42: Unknown | 2 | 1 | 0
  BILI, Day 42: Below | 0 | 0 | 0
  BILI, Day 42: Within | 50 | 55 | 90
  BILI, Day 42: Above | 0 | 0 | 3
  CREA, Day 0: number analyzed (Participants) | 30 | 38 | 59
  CREA, Day 0: Unknown | 0 | 0 | 0
  CREA, Day 0: Below | 1 | 0 | 1
  CREA, Day 0: Within | 28 | 33 | 54
  CREA, Day 0: Above | 1 | 5 | 4
  CREA, Day 21: Unknown | 1 | 0 | 2
  CREA, Day 21: Below | 7 | 2 | 1
  CREA, Day 21: Within | 44 | 53 | 90
  CREA, Day 21: Above | 1 | 2 | 4
  CREA, Day 42: number analyzed (Participants) | 52 | 56 | 93
  CREA, Day 42: Unknown | 2 | 1 | 0
  CREA, Day 42: Below | 5 | 2 | 2
  CREA, Day 42: Within | 45 | 52 | 85
  CREA, Day 42: Above | 0 | 1 | 6
  BUN, Day 0: number analyzed (Participants) | 30 | 38 | 59
  BUN, Day 0: Unknown | 0 | 0 | 0
  BUN, Day 0: Below | 0 | 0 | 0
  BUN, Day 0: Within | 28 | 37 | 57
  BUN, Day 0: Above | 2 | 1 | 2
  BUN, Day 21: Unknown | 1 | 0 | 2
  BUN, Day 21: Below | 1 | 0 | 0
  BUN, Day 21: Within | 49 | 52 | 92
  BUN, Day 21: Above | 2 | 5 | 3
  BUN, Day 42: number analyzed (Participants) | 52 | 56 | 93
  BUN, Day 42: Unknown | 2 | 1 | 0
  BUN, Day 42: Below | 0 | 0 | 0
  BUN, Day 42: Within | 47 | 47 | 89
  BUN, Day 42: Above | 3 | 8 | 4

25. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up period after the first vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 100
Participants
  Any AE(s) | 29 | 22 | 30
  Grade 3 AE(s) | 4 | 2 | 1
  Related AE(s) | 2 | 4 | 6

26. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: as for outcome 25
Time Frame: During the 83-day (Days 0-82) follow-up period after the first vaccination and the 62-day (Days 0-61) follow-up period after the second vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 100
Participants
  Any AE(s) | 37 | 26 | 41
  Grade 3 AE(s) | 8 | 4 | 7
  Related AE(s) | 2 | 4 | 6

27. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Month 12)
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
Number analyzed (Participants) | 53 | 57 | 100
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events (AEs): during the 21-day (Days 0-20) period after the first vaccination and 62-day (Days 0-61) period after the second vaccination; Serious adverse events (SAEs): during the entire study period (from Day 0 up to Month 12).
Arm/Group | GSK2340272A (3-5Y) Group | GSK2340272A (6-9Y) Group | GSK2340272A (10-17Y) Group
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/57 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/57 | 1/100
Other Adverse Events (participants affected / at risk) | 52/53 | 57/57 | 95/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A (3-5Y) Group (N=53) | GSK2340272A (6-9Y) Group (N=57) | GSK2340272A (10-17Y) Group (N=100)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2340272A (3-5Y) Group (N=53) | GSK2340272A (6-9Y) Group (N=57) | GSK2340272A (10-17Y) Group (N=100)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 20 (23) | 44 (60)
Chills (General disorders) | 11 (11) | 19 (21) | 38 (47)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 3 (3) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 28 (35) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 4 (5) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 22 (33) | 22 (33) | 33 (47)
Fatigue (General disorders) | 0 (0) | 35 (50) | 63 (95)
Gastroenteritis (Infections and infestations) | 4 (5) | 1 (1) | 3 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 17 (22) | 16 (23)
Headache (Nervous system disorders) | 3 (3) | 34 (51) | 71 (105)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 10 (10) | 9 (9) | 14 (16)
Irritability (Psychiatric disorders) | 21 (29) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 6 (6) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 23 (31) | 56 (82)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Otitis media (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 47 (85) | 56 (109) | 95 (181)
Pharyngitis (Infections and infestations) | 5 (6) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 34 (44) | 28 (34) | 34 (41)
Somnolence (Nervous system disorders) | 22 (28) | 0 (0) | 0 (0)
Swelling (General disorders) | 25 (34) | 30 (42) | 60 (91)
Tonsillitis (Infections and infestations) | 3 (3) | 1 (1) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 11 (15) | 3 (3) | 14 (19)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.